CLINICAL TRIAL: NCT04171752
Title: Open-label, Phase 1, Single-dose Study to Evaluate the Pharmacokinetics of Elafibranor 120 mg in Healthy Elderly and Young Adults Volunteers
Brief Title: Elafibranor Pharmacokinetic Parameters in Elderly Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GFT505-119-16; 2019-001819-23 (EudraCT Number)
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Geriatrics; Healthy
Keywords: elafibranor
MeSH Terms: interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, single-center, single-dose, two arms Phase 1 study in healthy elderly, aged of at least 75 years old (inclusive) and in healthy young adults, aged between 18 and 45 years old (all inclusive)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young Adults (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: elafibranor
- Elderly (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: elafibranor

INTERVENTIONS:
Drug: elafibranor — elafibranor 120mg is a coated tablet for oral administration
  Other Names: GFT505

SUMMARY:
In the elderly, pharmacokinetics is altered. Gastric juice pH is elevated which influences drug solubility and absorption. Drug distribution is decreased in the elderly because of decreased cardiac output, increased peripheral vascular resistance, diminished blood flow in the liver and the kidneys, reduced total amount of water in the body. Drug metabolism and biotransformation mainly take place in the liver and is often reduced. Drug elimination is altered very often because of reduced excretory (renal and hepatic) function. All these changes may lead to significant pharmacokinetic changes in geriatric population. A formal pharmacokinetic clinical study is being conducted in order to assess the need of dose adjustment in the elderly population.

ELIGIBILITY:
Inclusion Criteria:

- For All Participants:

1. Provide written informed consent prior to the conduct of any study related procedures;
2. With a minimum body weight (BW) of 50 kg and within a Body Mass Index (BMI) range of 18.0 to 30.0 kg/m^2 (all inclusive) at Screening visit;
3. Medically healthy as determined by the Investigator or medically qualified designee at both Screening and Inclusion visits. This will include no variation of BW of more than 5 percent between Screening and Inclusion visits;
4. Absence of clinically relevant abnormalities identified by a detailed medical history and complete physical examination;
5. Healthy participants, as determined by Normal Blood Pressure (BP) and Heart Rate (HR) at the screening and Inclusion visits after 5 minutes in supine position;
6. Normal ECG recording on a 12-lead ECG at the screening and Inclusion visits and no sign of any trouble of sinusal automatism, or considered as non clinically significant by investigator;
7. Laboratory parameters within the normal range of the laboratory;
8. Able to comprehend and willing to sign an Informed Consent Form, and to abide by the study restrictions;
9. Non-smoker participant or smoker of not more than 5 cigarettes/day within 3 months prior to Inclusion visit, and able to restrain from smoking during the whole study duration;
10. Participant with normal dietary habits;
11. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research;

    * For Healthy Young Volunteers only:
12. Males or females, between 18 and 45 years of age (all inclusive) at screening;
13. Matched to healthy elderly participants by BMI (plus or minus 20 percent) and gender;
14. Females participating in this study must be of non-childbearing potential or using highly efficient contraception for the full duration of the study and for 1 month after the end of treatment;
15. Females of childbearing potential must have a negative qualitative serum pregnancy test at Screening visit and a negative urine pregnancy test at Inclusion visit;

    * For Elderly volunteers only:
16. Males or females aged 75 years old or older at Screening visit;
17. Participants with mild, chronic, stable disease and stable treatment dose - no change in dose for the 3 months prior to Screening visit - (hypertension, hyperlipidemia, osteoarthritis, treated benign prostate hypertrophy, stable and treated hypothyroidism, treated glaucoma);
18. Participants with suitable veins for cannulation or repeated venipuncture.

Exclusion Criteria:

- For all participants:

1. Participants with a history of noncompliance to medical regimens;
2. Participant who, in the opinion of the Investigator, is likely to be not respectful or not cooperative during the study, or unable to cooperate because of a language problem or a mental deficiency;
3. Participant who cannot be contacted in case of emergency;
4. Participant who is in the exclusion period of a previous study;
5. Administrative or legal supervision;
6. Inability to abstain from intensive muscular effort;
7. Participant who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study;
8. A positive alcohol test result or urine screen for drugs of abuse result at Screening or Inclusion visits;
9. Any history or suspicion of alcohol abuse;
10. Any history or suspicion of consumption of any drug of abuse (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methamphetamines, methadone, methylenedioxymethamphetamine, opiates, tricyclic antidepressant), from screening to end of the study;
11. Consumption of nutritional supplements, herb-containing drug preparations (including Chinese medicines) or other foods or beverages (e.g., grapefruit and xanthine-containing foods or beverages) that may affect drug-metabolizing enzymes or transporters from screening to end of the study visit;
12. Evidence or history of gastrointestinal, hepatic, or renal disease, surgery or resection that would potentially alter absorption, distribution, metabolism, or excretion of orally administered drugs;
13. Participants who have clinically significant disease of cardiovascular, respiratory, renal, endocrine, hematological, gastrointestinal, neurological (central nervous system), psychiatric, systemic, infectious disorders or malignant tumor;
14. General anesthesia within 3 months before administration;
15. History or presence of allergy or unusual reactions to some drugs or anesthetics or known hypersensibility to the investigation product or its excipients;
16. Major surgery within 28 days prior to Screening visit or major surgery planned within 6 months following participation to the study;
17. Blood donation within 2 months before administration or blood donation planned during the study or within 2 months following participation to the study;
18. Receipt of blood products within 2 months prior to Inclusion visit;
19. Participants with symptomatic hypotension at Screening visit, whatever the decrease of blood pressure, or asymptomatic postural hypotension defined by a decrease in SBP ≥ 20 mmHg or DBP ≥ 10 mmHg within 3 minutes when changing from the supine to the standing position;
20. Frequent headaches and/or migraines, recurrent nausea and/or vomiting;
21. Participants who are positive for human immunodeficiency virus antibody, hepatitis B virus surface antigen, hepatitis C virus antibody;
22. Significant, uncontrolled, or life-threatening condition or organ or disease;
23. Show evidence of active renal disease (e.g. diabetic renal disease, polycystic kidney disease) or estimated glomerular filtration rate <60 mL/min/1.73m²;
24. Evidence of pelvic organ prolapsed, incontinence, or fistula of the urogenital system;
25. Have a history of syncope, presyncope, uncontrolled vertigo, postural dizziness, or at risk for falls, as judged to be clinically significant by the investigator;
26. Any drug intake during the 2 weeks or 5 half-life of the drug preceding the first administration except those defined in concomitant medication section

    * For Young Adults Volunteers only:
27. Females who are pregnant or breastfeeding. Female participants should not be enrolled if they plan to become pregnant during the time of study participation;
28. Any medications (except paracetamol 3g/day or contraception) intake within the 2 weeks or 5 half-life prior to Screening visit;
29. Evidence or history of clinically significant metabolic or allergic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics: Area under curve from dosing time to infinity (AUC(0-∞)) of elafibranor and active metabolite | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  In Healthy Young Adults compared to Healthy Elderly
Plasma pharmacokinetics: Area under curve from dosing time to last measurement (AUC(0-t)) of elafibranor and active metabolite | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  In Healthy Young Adults compared to Healthy Elderly
Plasma pharmacokinetics: maximum plasma drug concentration (Cmax) of elafibranor and active metabolite | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  In Healthy Young Adults compared to Healthy Elderly

SECONDARY OUTCOMES:
Plasma pharmacokinetics: elimination half-life (t1/2) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For elafibranor and metabolites
Plasma pharmacokinetics: area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total area under the plasma | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For elafibranor and metabolites
Plasma pharmacokinetics: time of maximum observed concentration (tmax) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For elafibranor and metabolites
Plasma pharmacokinetics: maximum plasma drug concentration (Cmax) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For other metabolites
Plasma pharmacokinetics: Area under curve from dosing time to infinity (AUC(0-∞)) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For other metabolites
Plasma pharmacokinetics: Area under curve from dosing time to last measurement (AUC(0-t)) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For other metabolites
Plasma pharmacokinetics: apparent volume of distribution (Vd/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For elafibranor
Plasma pharmacokinetics: renal clearance (CLr) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For elafibranor
Plasma pharmacokinetics: apparent non renal clearance (CLnr/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for elderly volunteers
  For elafibranor
Urine pharmacokinetics: amount excreted (Ae) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: cumulative amount excreted (Ae0-t) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: percentage of dose excreted (Fe) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: cumulative percent of dose excreted (Fe0-t) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: renal clearance (CLR) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Birman, MD, Study Director — Genfit
Locations (1):
- BIOTRIAL, Rennes, France

IPD SHARING:
Plan to Share IPD: No